CLINICAL TRIAL: NCT06063863
Title: Feasibility of Nurse-led Retinal Imaging for Retinopathy of Prematurity Screening Employing the Optos California
Acronym: N_ORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20046
Record Dates: First submitted 2023-07-20; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Retinopathy of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse led screening for ROP with OPTOS camera (Experimental): Screening completed by nurse trained in the use of an OPTOS camera to obtain images, at the same time as screening via standard procedure by a trained ophthalmologist using binocular indirect ophthalmoscopy (BIO).
  Interventions: Diagnostic Test: Nurse led screening with Optos ultra-widefield retinal-imaging device

INTERVENTIONS:
Diagnostic Test: Nurse led screening with Optos ultra-widefield retinal-imaging device — The screening will be completed by nurse trained in using an OPTOS camera, at the same time as screening for ROP by a trained ophthalmologist using standard procedure for screening for ROP using binocular indirect ophthalmoscopy (BIO). Images taken with OPTOS will then be remotely assessed by a qualified independent opthalmologist, to see if they can diagnose and grade ROP accurately using these images

SUMMARY:
Retinopathy of prematurity (ROP) is a preventable cause of blindness in babies who are born early i.e. premature. Internationally, there is a shortage of skilled ophthalmologists willing and able to screen for ROP. Even in the UK, not all hospitals have skilled ophthalmologists and premature babies have to travel to other hospitals, often long distances, to have their eyes examined. As a missed examination can lead to sight loss, this is a burden for families and carers of premature babies. To fill this gap, previous studies have explored the use of non-ophthalmologists healthcare workers to increase the workforce screening for ROP.

Recently, the Optos ultra-widefield retinal-imaging device (Optos PLC, Dunfermline, Scotland, UK) has been used to help document different stages of ROP in infants. This specialised retinal imaging system uses an internal ellipsoid mirror to capture fundal imaging angles of up to 200 degrees, or more than 80% of the entire retina, in a single image. A single retinal image can be acquired in a quarter of a second and is automatically captured when the infant's pupils are aligned with the Optos imaging device. No contact with the eye is necessary to capture an image of the retina. To date, there are no studies that have validated the Optos as a nurse-led screening tool for ROP.

This is a prospective study to determine and validate the feasibility of neonatal nurse-led retinal imagers for ROP screening employing the Optos imaging device. The main purpose of this study will be to test if it is possible for trained nurses to take good images of the back of babies eyes (retina) and if these images can be used by remotely placed ophthalmologists to diagnose and grade ROP. The investigators will compare how good the diagnosis and grading done using Optos images are compared to the current gold standard method (BIO). The investigators will also test how much agreement there is between ophthalmologists in interpreting Optos images by asking two ophthalmologists to grade the images.

DETAILED DESCRIPTION:
Retinopathy of Prematurity (ROP) is the major cause of blindness in babies who are born early i.e. premature (defined as those born at less than 37 weeks' gestation). All premature infants are at risk of developing ROP and are therefore routinely screened for the condition. With improvements, it has become one of the few preventable causes of childhood blindness, and recent reports suggest that most babies are saved from sight loss with proper screening and treatment. As neonatal care gets better, more premature babies are surviving and the need for ROP screening is increasing all over the world: about 8200 babies need screening in the UK each year. Very few babies need treatment - less than 2% in the UK. At the Royal Derby Hospital (RDH), about 4 to 5 infants are screened each week, with only 1 to 2 needing treatment per year.

The international classification of ROP describes ROP by its severity or stage (Stages 1-5), location by zone (I-III), extent by clock hours, and by the presence of pre-plus and plus disease. The aim of screening is to find out if the baby has any of these so that treatment can be done if needed. All babies born before 32 weeks or at less than 1500 g birth weight must have regular screening. For those born at <27 weeks gestation, the first ROP screening examination should be undertaken when at 30 to 31 weeks corrected gestational age while for babies who are more mature at birth, it is done between 4 to 5 weeks of actual age. Follow-up examinations should be performed every 1 to 2 weeks thereafter until the ophthalmologists (eye doctors) can see that the retina is fully matured. If there are signs of ROP, examinations should be performed more frequently, either weekly or twice a week.

All ROP screening examinations are currently done by a highly trained ophthalmologist using binocular indirect ophthalmoscopy (BIO), which is considered the gold standard method. The retinal findings are seen and drawn by hand in the patient's notes. These screening examinations are time-consuming for the ophthalmologist, and costly for the medical system as they need the ophthalmologist to be physically present and to do the screening. This makes it difficult for babies in remote hospitals or settings without trained ophthalmologists to have ROP screening. To reduce this difficulty several groups have developed cameras that can take pictures of the retina. The pictures can then be transferred to ophthalmologists who can diagnose and grade the ROP remotely.

The most common imaging system used for ROP screening is the RetCam (Clarity Medical Systems, Pleasanton, California, USA). The RetCam imaging system, a hand-held camera, is connected by a fiber optic cable to an electro-optical box housed in a movable cart. To take images with RetCam, the babies pupils have to be dilated (opened up) by using medicines and local painkillers. The eyelids are held open with a lid speculum and the camera probe is applied with a contact lens gel such that it is touching the front of the eye, over the open pupil. RetCam images are not able to include the whole of the back of the eye in one picture and therefore multiple images have to be taken. This takes time and effort from highly-skilled imagers. Also, the picture quality is not good if the pupil is not opened properly or if there is some obstruction in the way such as blood in the eye. As the camera has to touch the eye, it can hurt the eye and make the baby uncomfortable such as by stimulating eye nerves that cause the heart to slow down and lower the baby's blood oxygen levels. Too much pressure on the eye can also change the picture and make the diagnosis difficult.

More recently, a new camera, the Optos ultra-widefield retinal-imaging device (Optos PLC, Dunfermline, Scotland, UK) has been used to take and store pictures of different stages of ROP in babies. This camera has a specialised mirror to capture pictures that contain details of nearly all of the retina in a single photo. It is quick, the complete single photo can the taken in a quarter of a second. In addition, it can take pictures without touching the baby's eyes so there is no risk of damage to the eye. Thus, the Optos camera has many advantages over the RetCam.

If this camera could be used by nurses trained to take pictures and ophthalmologists could diagnose and grade ROP from these pictures, babies could be screened without every hospital needing to have a specially trained ophthalmologist or the baby travelling distances to go to a centre that had such a doctor. As most babies only need screening, ophthalmologists could ask for only those who need treatment (about 2 in 100 babies) to be transferred to specialist centres. This could reduce the cost of care to the NHS and problems for families of premature babies.

In the Derby neonatal unit, the study team have already tested the Optos camera and found that it is safe to use in babies and did not cause them any undue discomfort. In this study, the study team want to see if it is possible to train a nurse to take pictures of the retina using the Optos camera and if ophthalmologists can diagnose and grade ROP accurately using these images. No studies have been done to test this.

ELIGIBILITY:
Inclusion Criteria:

* Infants (upper age limit 1 years old) eligible for routine ROP screening as part UK ROP screening guidelines (any infant born at or before 32 weeks' gestation and / or weigh 1500 grams or less).
* Infants with parents/legal guardians who can give written informed consent.

Exclusion Criteria:

* Infants not eligible for routine ROP screening under UK ROP screening guidelines.
* Infants who are deemed not well enough by the attending consultant neonatologist for retinal examination or retinal imaging.
* Any premature infant with media opacities that prevents adequate visualisation of the retina.
* Inability of the parents to give written, informed consent.

Ages: 32 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Retinopathy of prematurity diagnosis | 18 months
  To evaluate the agreement by measuring the Kappa Co-efficient for agreement, for diagnosis and grading of ROP and posterior pole (pre-plus or plus disease) and peripheral retinal vascular changes, between nurse-led OPTOS imaging and indirect Ophthalmoscopy performed by an ophthalmologist.
Retinopathy of prematurity grading | 18 months
  To evaluate the agreement by measuring the Kappa Co-efficient for agreement, for diagnosis and grading of ROP and posterior pole (pre-plus or plus disease) and peripheral retinal vascular changes, between nurse-led OPTOS imaging and indirect Ophthalmoscopy performed

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Ojha, Professor, Principal Investigator — University of Nottingham
Locations (1):
- University Hospitals of Derby and Burton, Derby, Derbyshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fung THM, Abramson J, Ojha S, Holden R. Systemic Effects of Optos versus Indirect Ophthalmoscopy for Retinopathy of Prematurity Screening. Ophthalmology. 2018 Nov;125(11):1829-1832. doi: 10.1016/j.ophtha.2018.06.001. Epub 2018 Jul 6. No abstract available. PMID 30322451